CLINICAL TRIAL: NCT05678088
Title: Strengthening Oropharyngeal Muscles as a Novel Approach to Treat Obstructive Sleep Apnea: A Randomized Feasibility Study
Brief Title: Oropharyngeal Exercises to Treat Obstructive Sleep Apnea
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Mark Boulos, MD, Principal Investigator, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5541
Record Dates: First submitted 2022-12-15; First posted 2023-01-10 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; Oropharyngeal Exercises
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Supervised Oropharyngeal Exercises (Experimental): The participant will perform the oropharyngeal exercises that strengthen the tongue and pharyngeal muscles. The protocol will be delivered via a tablet-based app. The speech language pathologist will call or conduct videoconference visits with participants 1, 3, 5, 7 and 9 weeks after the baseline assessment to provide re-training (if needed) and to troubleshoot technical issues related to the use of the app.
  Interventions: Behavioral: Oropharyngeal Exercises
- Unsupervised Oropharyngeal Exercises (Active Comparator): The participant will perform the oropharyngeal exercises that strengthen the tongue and pharyngeal muscles. The protocol will be delivered via a tablet-based app. After the initial training there will be no further scheduled interactions with the study staff except during the follow-up telephone calls and study visits.
  Interventions: Behavioral: Oropharyngeal Exercises
- Supervised Sham Exercises (Sham Comparator): The participant will perform sham control exercises that have no impact on oropharyngeal (e.g., base of the tongue) muscle strength. The speech language pathologist will call or conduct videoconference visits with participants 1, 3, 5, 7 and 9 weeks after the baseline assessment to provide re-training (if needed) and to troubleshoot technical issues related to the use of the app.
  Interventions: Behavioral: Sham Exercises

INTERVENTIONS:
Behavioral: Oropharyngeal Exercises — The participant will practice exercises designed to strengthen the tongue and pharyngeal muscles
  Arms: Supervised Oropharyngeal Exercises; Unsupervised Oropharyngeal Exercises
Behavioral: Sham Exercises — The participant will practice exercises that have no impact on oropharyngeal (e.g., base of the tongue) muscle strength.
  Arms: Supervised Sham Exercises

SUMMARY:
The goal of this study is to determine whether a randomized controlled trial using oropharyngeal exercises to treat sleep apnea is feasible. Continuous positive airway pressure (CPAP) is the standard therapy for Obstructive sleep apnea (OSA), but it is poorly tolerated by many patients. Oropharyngeal exercises (OPEs) which are commonly used by speech-language pathologists to improve oro-motor strength, may serve as a promising alternative approach. The main questions this study aims to answer are:

* Is it feasible to use an oropharyngeal exercise protocol in patients with sleep apnea?
* Will oropharyngeal exercises improve sleep apnea severity, daytime sleepiness, sleep quality, mood, workplace performance, and quality of life

Participants will be randomized into a supervised OPE intervention arm vs. unsupervised OPE intervention arm vs. sham treatment for a 10-week/5-day per week/two 20-minute session exercise protocol. The exercises will be administered via an app and the investigators will assess feasibility, as well as several sleep-related and oro-motor physiological outcomes before treatment, immediately post-treatment, and 4 weeks post-treatment. The investigators will use the results of this feasibility trial to inform the sample size needed for a larger clinical trial that will determine the efficacy of using oropharyngeal exercises to treat OSA.

DETAILED DESCRIPTION:
1. BACKGROUND

   Obstructive sleep apnea (OSA) is a common disorder, and it is estimated that approximately one third of adult Canadians are at risk for obstructive sleep apnea (OSA), and approximately 20% of the general population has been diagnosed with OSA. Few effective treatment options are available to individuals with OSA. Continuous positive airway pressure (CPAP) is first-line therapy for treating moderate to severe OSA, and acts as a pneumatic splint to keep the airway open during sleep. Although CPAP is generally effective at treating OSA, it remains poorly tolerated by many patients; rates of non-adherence are estimated to be as high as 46 to 83%, with only one third of patients using CPAP at 4 years.

   Oropharyngeal exercises (OPEs) are commonly used by speech-language pathologists to improve oro-motor strength and range of motion and serve as a promising alternative approach to treat OSA. Studies conducted so far have demonstrated that oropharyngeal exercises may be beneficial in the treatment of OSA. However, two recent systematic reviews concluded that the quality of the available evidence was low and larger blinded studies were needed.
2. RATIONALE

   Due to poor rates of adherence, there is a major clinical need to develop alternative treatments to CPAP for OSA that are effective and well-tolerated. While oropharyngeal exercises appear to be a highly promising alternative approach to treat OSA, their efficacy in reducing OSA severity has not been established, and feasibility of this approach has not been demonstrated.
3. STUDY GOALS

   Research Question: Is a randomized controlled trial (RCT) of an oropharyngeal exercise regimen in patients with OSA feasible?

   Primary Objective: The investigators will determine the feasibility of a randomized controlled trial of an oropharyngeal exercise regimen (involving supervised vs. unsupervised exercises) in patients with moderate to severe OSA who cannot tolerate or are unwilling to use CPAP. The investigators will assess the following: (i) rate of recruitment (ii) adherence to the study exercise intervention. (iii) Ability to ascertain OSA severity (which will be the primary outcome for the full trial).

   Secondary Objectives: The investigators will secondarily obtain refined estimates of variability around OSA severity, daytime sleepiness, sleep quality, mood, workplace performance, and quality of life. This will help refine the sample size estimate for the subsequent trial. Furthermore, the investigators will assess the acceptability, appropriateness, and feasibility of the intervention from the perspective of the participants.
4. SIGNIFICANCE

Untreated OSA is a hidden healthcare crisis associated with numerous adverse health and economic consequences. If oropharyngeal exercises are found to be efficacious for the management of OSA, this would provide a novel low-cost, non-pharmacological treatment for OSA that could address current undertreatment due to socioeconomic factors and poor patient tolerance. The proposed feasibility study is the first step to demonstrating potential efficacy of this intervention in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patients with OSA (defined as an apnea-hypopnea index ≥10/hr) in whom >50% of the respiratory events are obstructive in nature
* Patients who are unwilling to use CPAP or have been unable to tolerate CPAP after at least a 2-week trial
* Patients who are also not using an equipment-based treatment modality (e.g. PAP therapy, a dental appliance, or hypoglossal nerve stimulation) or surgery to manage their OSA.

Exclusion Criteria:

* Planned airway surgery, use of CPAP, a dental appliance, or other equipment-based treatment modality to manage OSA during the course of the study
* Central respiratory events account for ≥50% of the overall apnea-hypopnea index
* Reduced cognition (MoCA<18)
* Any significant neurological condition that could impact oropharyngeal activity
* Use of medications that may impact tone of the upper airway (e.g. hypnotics, opiates) ≥3 nights per week during the 4 weeks prior to randomization
* Use of a medical device that would interfere with the use of the home sleep apnea test
* Plans to move to another city during the study that would impact compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-03-28 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Rate of recruitment | 2 years
  The study team will maintain logs to track the number of patients screened, found to be eligible, and randomized into the trial; we will also track dropouts
Patient adherence with the study exercises | 10 weeks
  Patient adherence with the study exercises will be tracked (in minutes) by the OPEX app that will deliver the oropharyngeal/sham exercises. We will compute the percentage of exercises completed.
Ability to ascertain Obstructive Sleep Apnea (OSA) severity | 14 weeks
  Ability to ascertain OSA severity, as assessed by completion rates for the three home sleep apnea tests at baseline, post-training and retention. A home sleep apnea test will be considered "completed" if ≥4 hours of flow, effort, and oxygen evaluation are obtained. The cut-off of ≥4 hours was selected as it has been recommended by clinical practice guidelines and previously used in prior home sleep apnea test feasibility studies.

SECONDARY OUTCOMES:
Change in Obstructive Sleep Apnea (OSA) Severity (as measured by the apnea-hypopnea index) | Baseline to 10 weeks (post-training) and 14 weeks (retention)
  Measured by the apnea-hypopnea index (AHI). AHI quantifies the number of apneas and hypopneas per hour of sleep. It will be measured using a home sleep monitor.
Change in Lowest Oxygen Desaturation | Baseline to 10 weeks (post-training) and 14 weeks (retention)
  Lowest oxygen desaturation will be measured using a home sleep monitor.
Change in Objective sleep quality | Baseline to 10 weeks (post-training) and 14 weeks (retention)
  Objective sleep quality and quantity will be assessed using wrist actigraphy that will be provided with the home sleep apnea test. Sleep efficiency will be calculated by dividing the amount of time spent asleep (in minutes) by the total amount of time in bed (in minutes).
Change in Objective sleep quantity | Baseline to 10 weeks (post-training) and 14 weeks (retention)
  Objective sleep quality will be assessed using wrist actigraphy that will be provided with the home sleep apnea test. The total sleep time will be calculated.
Change in Sleep Quality (as assessed by the Pittsburgh Sleep Quality Index) | Baseline to 2 weeks, 6 weeks, 10 weeks (post-training), 12 weeks, 14 weeks (retention)
  Sleep quality as assessed by the Pittsburgh Sleep Quality Index. The questionnaire is scored on a range from 0-21 points, with "0" indicating no difficulty and "21" indicating severe difficulties in all areas.
Change in Daytime Sleepiness (as assessed by the Epworth Sleepiness Scale) | Baseline to 2 weeks, 6 weeks, 10 weeks (post-training), 12 weeks, 14 weeks (retention)
  Scores on Epworth Sleepiness Scale range from range from 0 to 24, with higher scores indicating higher average sleep propensity in daily life (daytime sleepiness).
Change in Mood (as assessed by the Beck Depression Inventory) | Baseline to 2 weeks, 6 weeks, 10 weeks (post-training), 12 weeks, 14 weeks (retention)
  The Beck Depression Inventory has 21 questions that are scored on a range of 0-63 points. Higher scores indicate more severe depression.
Change in Workplace performance (as assessed by the Work Limitations Questionnaire) | Baseline to 2 weeks, 6 weeks, 10 weeks (post-training), 12 weeks, 14 weeks (retention)
  Workplace performance as assessed by the Work Limitations Questionnaire. There are 25 items, that address 4 scales: Time Management, Physical Demands, Mental-Interpersonal Demands, and Output Demands. Scale scores range from 0 (limited none of the time) to 100 (limited all of the time) and represent the reported amount of time in the prior two weeks respondents were limited on-the-job.
Change in Self-reported Quality of Life as assessed by the EQ-5D-5L | Baseline to 2 weeks, 6 weeks, 10 weeks (post-training), 12 weeks, 14 weeks (retention)
  The EQ-5D-5L questionnaire has 5 dimensions: Mobility, Self-Care, Usual Activity, Pain/Discomfort, Anxiety/Depression, with each dimension rated on a level from 1-5 where higher scores indicate more severe problems.
Change in Self-reported Quality of Life (as assessed by the SF-36 Questionnaire) | Baseline to 2 weeks, 6 weeks, 10 weeks (post-training), 12 weeks, 14 weeks (retention)
  The SF-36 Questionnaire has 36-items that covers eight areas: physical functioning, bodily pai, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. Scores for each domain range from 0 to 100, with a higher score indicating better health.
Acceptability, Appropriateness, and Feasibility of Intervention Measure | 10 weeks
  Acceptability, Appropriateness, and Feasibility of Intervention Measure Questionnaire contains 4 questions for each dimension (acceptability, appropriateness, and feasibility). Each question is rated from 1-5, and higher scores indicate that participants believe this is a more acceptable, appropriate, or feasibly intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Boulos, MD, MSc, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Epstein LJ, Kristo D, Strollo PJ Jr, Friedman N, Malhotra A, Patil SP, Ramar K, Rogers R, Schwab RJ, Weaver EM, Weinstein MD; Adult Obstructive Sleep Apnea Task Force of the American Academy of Sleep Medicine. Clinical guideline for the evaluation, management and long-term care of obstructive sleep apnea in adults. J Clin Sleep Med. 2009 Jun 15;5(3):263-76. PMID 19960649
- [Background] Weaver TE, Grunstein RR. Adherence to continuous positive airway pressure therapy: the challenge to effective treatment. Proc Am Thorac Soc. 2008 Feb 15;5(2):173-8. doi: 10.1513/pats.200708-119MG. PMID 18250209
- [Background] Hsu B, Emperumal CP, Grbach VX, Padilla M, Enciso R. Effects of respiratory muscle therapy on obstructive sleep apnea: a systematic review and meta-analysis. J Clin Sleep Med. 2020 May 15;16(5):785-801. doi: 10.5664/jcsm.8318. Epub 2020 Feb 6. PMID 32026802
- [Background] Rueda JR, Mugueta-Aguinaga I, Vilaro J, Rueda-Etxebarria M. Myofunctional therapy (oropharyngeal exercises) for obstructive sleep apnoea. Cochrane Database Syst Rev. 2020 Nov 3;11(11):CD013449. doi: 10.1002/14651858.CD013449.pub2. PMID 33141943
- [Background] Franklin KA, Lindberg E. Obstructive sleep apnea is a common disorder in the population-a review on the epidemiology of sleep apnea. J Thorac Dis. 2015 Aug;7(8):1311-22. doi: 10.3978/j.issn.2072-1439.2015.06.11. PMID 26380759